CLINICAL TRIAL: NCT07365813
Title: Developing and Testing AI-Generated Messages on Alcohol and Cancer Risk: A Proof of Concept
Brief Title: Testing Alcohol Cancer Risk Messages
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Taghrid Asfar, Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20250012
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Alcohol; Cancer
Keywords: alcohol; alcohol warning labels; cancer survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gain-framed Messages (Experimental): The study will test in an online 15 minutes single session, four gain-framed alcohol-cancer risk messages. Each message will be viewed in three intensity levels (text-only, neutral image, and graphic image), yielding 12 total message stimuli.
  Interventions: Behavioral: Text-only messages; Behavioral: AI-developed Neutral pictorial messages; Behavioral: AI-developed graphic pictorial messages
- Loss-Framed Messages (Experimental): The study will test in an online 15 minutes single session, four loss-framed alcohol-cancer risk messages. Each message will be viewed in three intensity levels (text-only, neutral image, and graphic image), yielding 12 total message stimuli.
  Interventions: Behavioral: Text-only messages; Behavioral: AI-developed Neutral pictorial messages; Behavioral: AI-developed graphic pictorial messages

INTERVENTIONS:
Behavioral: Text-only messages — The study will test eight alcohol-cancer risk messages (four gain-framed and four loss-framed). Each message will be developed at three intensity levels (text-only, neutral image, and graphic image), yielding 24 total message stimuli.
Behavioral: AI-developed Neutral pictorial messages — The study will test eight alcohol-cancer risk messages (four gain-framed and four loss-framed). Each message will be developed at three intensity levels (text-only, neutral image, and graphic image), yielding 24 total message stimuli.
Behavioral: AI-developed graphic pictorial messages — The study will test eight alcohol-cancer risk messages (four gain-framed and four loss-framed). Each message will be developed at three intensity levels (text-only, neutral image, and graphic image), yielding 24 total message stimuli.

SUMMARY:
Testing gain vs loss-framed messages to address drinking among cancer survivors

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Resident of the United States
* Able to read and speak English
* Diagnosed with one of the following cancers: mouth, throat, larynx, liver, colon, rectum, or breast
* Current alcohol user (≥ 1 alcoholic drink in the past 30 days)

Exclusion Criteria:

* Adults unable to consent
* Individuals younger than 21
* Not residing in the US
* Non-alcohol users (<1 drink)
* Less than 50% completion of the survey

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol-cancer harm perception | Within 15 minutes on a single online session - from before message exposure (pre-exposure) to after message exposure (post-exposure).
  Change in participants' beliefs about experiencing cancer in the future due to alcohol use measured on a scale from 1 (not at all) to 5 (a lot). The outcome is the change on the mean score from the pre to post exposure.
Intention to Reduce Alcohol consumption | Within 15 minutes on a single online session - from before message exposure (pre-exposure) to after message exposure (post-exposure).
  Change in participants' intention to reduce alcohol consumption in the next month, measured on a scale from 1 (not at all) to 5 (a lot). The outcome is the change on the mean score from the pre to post exposure.
Commitment to a limited drinking goal in the next month | Within 15 minutes on a single online session - from before message exposure (pre-exposure) to after message exposure (post-exposure).
  Change in participants' intention to commit to a drinking limit goal in the next month, measured on a scale from 1 (not at all) to 5 (a lot). The outcome is the change on the mean score from the pre to post exposure.

SECONDARY OUTCOMES:
Message perceived effectiveness | One time (within 5 minutes) post-exposure evaluation.
  Self reported perceived overall effectiveness of the message measured on a scale from 1 (not at all) to 5 (a lot) scale. The outcome is the mean score.
Message Receptivity | One time (within 5 minutes) post-exposure evaluation.
  Self reported message receptivity including attention, emotional reaction, believability, fear, relevance, anticipated social interactions, recall and avoidance on a scale from 1 (not at all) to 5 (a lot). The outcome is the composite mean score assessing attention, emotional reaction, believability, fear, relevance, anticipated social interactions, recall, avoidance, and perceived effectiveness. Higher scores indicate greater message receptivity.

CONTACTS AND LOCATIONS:
Overall Officials: Taghrid Asfar, MD, MSPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No